CLINICAL TRIAL: NCT06004570
Title: Effects of a Combination of Polyphenol-rich Extracts on the Protection of Retinal Cells Against Blue Light in the Prevention of Ocular Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AronPharma Sp. z o. o. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 05-AP-RET
Record Dates: First submitted 2023-08-07; First posted 2023-08-22 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-08

CONDITIONS: Eye Abnormalities
Keywords: Retinal cells; Ocular diseases; Blue-light
MeSH Terms: conditions — Eye Abnormalities

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Complex product (Experimental): 18 volunteers
  Interventions: Dietary Supplement: Complex product
- Polyphenol-rich extracts (Active Comparator): 18 volunteers
  Interventions: Dietary Supplement: Polyphenol-rich extracts
- Placebo (Placebo Comparator): 18 volunteers
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Complex product — Extracts from the fruits of Vaccinium myrtillus L. + Aronia Melanocarpa (Michx.) Elliot + Lonicera caerulea var. Kamtschatica, rutin, vitamin B6, vitamin B12, folic acid Single oral dose - 2 capsules
  Arms: Complex product
Dietary Supplement: Polyphenol-rich extracts — Extracts from the fruits of Vaccinium myrtillus L. + Aronia Melanocarpa (Michx.) Elliot + Lonicera caerulea var. Kamtschatica Single oral dose - 2 capsules
  Arms: Polyphenol-rich extracts
Other: Placebo — Single oral dose - 2 capsules
  Arms: Placebo

SUMMARY:
The aim of the study is to confirm that daily supplementation with a product containing a standardized combination of polyphenol-rich extracts has a protective effect against potential blue-light-induced damage to retinal cells.

DETAILED DESCRIPTION:
Randomized, double-blind, parallel study conducted under medical supervision on a group of 54 volunteers exposed to blue-light for 6-8h a day. Patients receive one of the investigational products or placebo for 6 weeks. Study parameters: OCT (optical coherence tomography), Amsler test, Computerized Perimetry, Schirmer test. In addition, subjective symptoms will be assessed using the Visual Analog Scale (VAS) method and a Dry Eye-Related Quality-of-Life Questionnaire. The studied parameters will be measured before and after supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Women and men, 25-45 years old.
* Signed informed consent.
* Volunteers who do not use glasses or contact lenses.
* Volunteers exposed to blue light for at least 6 - 8 hours a day.

Exclusion Criteria:

* Intake of supplements containing plant extracts, polyphenols or anthocyanins.
* Participation in another clinical trial.
* Oncological disease, autoimmune disease, severe liver dysfunction, tuberculosis, leukemia, multiple sclerosis, AIDS, rheumatoid arthritis, organ transplant and other gastrointestinal diseases that may affect the results of the study.
* Women who are pregnant, planning to become pregnant during the study, or breastfeeding.
* Use of drugs that cause impaired vision or impaired tear secretion (including digoxin, fluoroquinolones, metronidazole, hydrochlorothiazide, retinoids).
* Current use of eye drops in the treatment of ocular diseases.
* Ocular diseases.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
DEQS (Dry Eye-Related Quality-of-Life) index | Baseline, 6 weeks
  Subjective symptom questionnaire assessment
Visual Analogue Scale | Baseline, 6 weeks
  Subjective symptom assessment

SECONDARY OUTCOMES:
Optical Coherence Tomography | Baseline, 6 weeks
  An OCT provides cross sectional images of the retina to enable early detection and treatment of ocular disease
Amsler test | Baseline, 6 weeks
  Amsler grid usually help detecting defects in central 20 degrees of the visual field
Schirmer test, | Baseline, 6 weeks
  Schirmer test quantitatively measures the tear production by the lacrimal gland
Computerized Perimetry | Baseline, 6 weeks
  Computerized Perimetry is used to evaluate visual function

CONTACTS AND LOCATIONS:
Locations (1):
- Centrum Zdrowia Eter-Med sp. z o.o., Gdansk, Poland

IPD SHARING:
Plan to Share IPD: No